CLINICAL TRIAL: NCT04529759
Title: Tolerance of Healthy Term Infants Fed Milk-Based Infant Formula With Oligosaccharides
Brief Title: Healthy Term Infants Fed Milk-Based Infant Formula
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: AL39
Record Dates: First submitted 2020-08-25; First posted 2020-08-28 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2021-07

CONDITIONS: Tolerance

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Infant Formula (Active Comparator): Feed ad libitum
  Interventions: Other: Control Infant Formula
- Experimental Infant Formula (Experimental): Feed ad libitum
  Interventions: Other: Experimental Infant Formula

INTERVENTIONS:
Other: Control Infant Formula — Powdered partially hydrolyzed whey (WPH) based formula with an oligosaccharide
  Arms: Control Infant Formula
Other: Experimental Infant Formula — Powdered partially hydrolyzed whey (WPH) based formula with oligosaccharides blend
  Arms: Experimental Infant Formula

SUMMARY:
This is a randomized, controlled, double-blind, parallel, feeding study with the purpose to evaluate the tolerance of healthy term infants fed partially hydrolyzed whey protein infant formulas.

ELIGIBILITY:
Inclusion Criteria:

* Good health as determined from participant's medical history
* Singleton from a full-term birth with a gestational age of 37-42 weeks
* Birth weight was > 2490 g (~5 lbs. 8 oz.)
* Parent(s) confirm their intention to feed their infant the study product as the sole source of nutrition for the duration of the study
* Parent(s) confirm their intention not to administer vitamin or mineral supplements, (except for vitamin D supplements if instructed by their healthcare professional), solid foods or juices to their infant from enrollment through the duration of the study
* Participant's parent(s) has voluntarily signed and dated an Informed Consent Form (ICF), approved by an Institutional Review Board/Independent Ethics Committee (IRB/IEC) and provided Health Insurance Portability and Accountability Act (HIPAA) (or other applicable privacy regulation) authorization prior to any participation in the study

Exclusion Criteria:

* An adverse maternal, fetal or participant medical history that is thought by the investigator to have potential for effects on tolerance, growth, and/or development
* Participant is taking and plans to continue taking medications (including over the counter (OTC), such as Mylicon® for gas), prebiotics, probiotics, home remedies (such as juice for constipation), herbal preparations or rehydration fluids that might affect gastrointestinal (GI) tolerance
* Participant is enrolled in another study that has not been approved as a concomitant study

Max Age: 14 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 108 (Actual)
Dates: Start 2020-09-12 (Actual); Primary Completion 2021-06-18 (Actual); Study Completion 2021-06-18 (Actual)

PRIMARY OUTCOMES:
Mean rank stool consistency (MRSC) | Study Day 1 to 28 Days of Age
  Parent Completed Diary

SECONDARY OUTCOMES:
Weight | 14 to 119 Days of Age
  Interval weight gain per day
Gastrointestinal tolerance | 14 to 119 Days of Age
  Parent Completed Diary
Length | 14 to 119 Days of Age
  Interval length gain per day
Head Circumference | 14 to 119 Days of Age
  Interval head circumference gain per day

OTHER OUTCOMES:
Infant Stool Characteristics | Study Day 1 to 119 Days of Age
  Parent Completed Diary
Study Product Intake | Study Day 1 to 119 Days of Age
  Parent Completed Diary
Infant and Household Characteristics | Study Day 1 to 119 Days of Age
  Parent reported lifestyle and illness questions
Health Resource Utilization | Study Day 1 to 119 Days of Age
  Number of Visits
Infant Feeding and Stool Patterns Questionnaire | Exit or 119 Days of Age
  Parent completed questionnaire; 16, 5-point Likert scale questions, scaled in the negative direction
Infant Behavior Questionnaire | Exit or 119 Days of Age
  Parent completed questionnaire; 22 questions with 5-point Likert scale questions; scaled in the negative direction
Formula Satisfaction Questionnaire | Exit or 119 Days of Age
  Parent completed questionnaire; 13 questions of up to 5 categories scaled in the negative direction
Adverse Events | Study Day 1 to 119 Days of Age
  Standard adverse event reporting

CONTACTS AND LOCATIONS:
Overall Officials: John Lasekan, PhD, Study Chair — Abbott Nutrition
Locations (6):
- United States (6):
  - Visions Clinical Research, Tucson, Arizona
  - PAS Research, LLC, Tampa, Florida
  - Springs Medical Research, Owensboro, Kentucky
  - Institute of Clinical Research, Mentor, Ohio
  - The Cleveland Pediatric Research Center, LLC, Westlake, Ohio
  - Midsouth Center for Clinical Research, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No